CLINICAL TRIAL: NCT03770403
Title: A Long-Term, Single-Arm, Open-Label, Multicenter, Phase 3 Follow-on Trial of ARGX-113-1704 to Evaluate the Safety and Tolerability of ARGX-113 in Patients With Myasthenia Gravis Having Generalized Muscle Weakness
Brief Title: A Safety and Tolerability Study of ARGX-113 in Patients With Myasthenia Gravis Who Have Generalized Muscle Weakness.
Acronym: ADAPT+
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-1705; 2018-002133-37 (EudraCT Number)
Expanded Access: NCT04777734 (Approved for marketing)
Record Dates: First submitted 2018-11-16; First posted 2018-12-10 (Actual); Results first posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARGX-113 (Experimental)
  Interventions: Biological: ARGX-113

INTERVENTIONS:
Biological: ARGX-113 — Intravenous administration of ARGX-113
  Other Names: efgartigimod

SUMMARY:
This is a Long-Term, Single-Arm, Open-Label, Multicenter Phase 3 follow-on trial of the ARGX-113-1704 study to evaluate the safety and tolerability of ARGX-113 in patients with gMG. Patients who have completed at least 1 cycle of treatment and at least 1 year of trial ARGX-113-1705 and have started Part B are eligible to enroll in the open-label trial ARGX-113-2002 to receive efgartigimod by SC administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the ability to understand the requirements of the trial, provide written informed consent, and comply with the trial protocol procedures.
2. Patients who participated in trial ARGX-113-1704 and are eligible for roll over, as specified in the protocol.

Other more specific inclusion criteria are further defined in the protocol.

Exclusion Criteria:

1. Patients who discontinued early from trial ARGX-113-1704 or patients who discontinued early from randomized treatment for pregnancy or rescue reasons or an (S)AE that might jeopardize the safety of the patient in that trial.
2. Pregnant and lactating women, and those intending to become pregnant during the trial or within 90 days after the last dosing. Women or childbearing potential should have a negative urine pregnancy test at SEB.
3. Male patients who are sexually active and do not intend to use effective methods of contraception during the trial or within 90 days after the last dosing or male patients who plan to donate sperm during the trial or within 90 days after the last dosing.
4. Patients with known Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV) seropositivity.

Other, more specific exclusion criteria are further defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Coppieters, MD, Study Director — argenx
Locations (52):
- United States (14):
  - Investigator Site 42, Carlsbad, California
  - Investigator Site 8, Los Angeles, California
  - Investigator Site 33, Orange, California
  - Investigator Site 21, Palo Alto, California
  - Investigator Site 41, Jacksonville, Florida
  - Investigator Site 4, Tampa, Florida
  - Investigator Site 14, Kansas City, Kansas
  - Investigator Site 32, Detroit, Michigan
  - Investigator Site 2, Chapel Hill, North Carolina
  - Investigator Site 18, Cleveland, Ohio
  - Investigator Site 12, Portland, Oregon
  - Investigator Site 1, Cordova, Tennessee
  - Investigator Site 3, San Antonio, Texas
  - Investigator Site 37, Charlottesville, Virginia
- Belgium (2):
  - Investigator Site 11, Edegem
  - Investigator Site 7, Ghent
- Canada (2):
  - Investigator Site 20, Toronto, Ontario
  - Investigator Site 25, Montreal, Quebec
- Czechia (3):
  - Investigator Site 16, Brno
  - Investigator Site 19, Ostrava-Poruba
  - Investigator Site 30, Prague
- Denmark (2):
  - Investigator Site 49, Aarhus
  - Investigator Site 17, Copenhagen
- France (2):
  - Investigator Site 50, Bordeaux
  - Investigator Site 51, Marseille
- Georgia (3):
  - Investigator Site 45, Tbilisi
  - Investigator Site 31, Tbilisi
  - Investigator Site 46, Tbilisi
- Investigator Site 28, Berlin, Germany
- Hungary (2):
  - Investigator Site 35, Budapest
  - Investigator Site 52, Szeged
- Italy (3):
  - Investigator Site 10, Milan, MI
  - Investigator Site 5, Napoli
  - Investigator Site 38, Roma
- Japan (10):
  - Investigator Site 24, Sapporo, Hokkaido
  - Investigator Site 13, Hanamaki-shi, Iwate
  - Investigator Site 27, Sendai, Miyagi
  - Investigator Site 23, Ōsaka-sayama, Osaka
  - Investigator Site 22, Suita, Osaka
  - Investigator Site 40, Meguro City, Tokyo
  - Investigator Site 43, Shinjuku-Ku, Tokyo
  - Investigator Site 47, Chiba
  - Investigator Site 44, Hiroshima
  - Investigator Site 48, Minato
- Investigator Site 36, Leiden, Netherlands
- Poland (4):
  - Investigator Site 9, Gdansk
  - Investigator Site 29, Katowice
  - Investigator Site 6, Krakow
  - Investigator Site 15, Warsaw
- Russia (2):
  - Investigator Site 34, Novosibirsk
  - Investigator Site 39, Samara
- Investigator Site 26, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howard JF Jr, Bril V, Vu T, Karam C, Peric S, De Bleecker JL, Murai H, Meisel A, Beydoun SR, Pasnoor M, Guglietta A, Van Hoorick B, Steeland S, T'joen C, Utsugisawa K, Verschuuren J, Mantegazza R; ADAPT+ Study Group. Long-term safety, tolerability, and efficacy of efgartigimod (ADAPT+): interim results from a phase 3 open-label extension study in participants with generalized myasthenia gravis. Front Neurol. 2024 Jan 17;14:1284444. doi: 10.3389/fneur.2023.1284444. eCollection 2023. PMID 38318236
- [Derived] Howard JF Jr, Bril V, Vu T, Karam C, Peric S, Margania T, Murai H, Bilinska M, Shakarishvili R, Smilowski M, Guglietta A, Ulrichts P, Vangeneugden T, Utsugisawa K, Verschuuren J, Mantegazza R; ADAPT Investigator Study Group. Safety, efficacy, and tolerability of efgartigimod in patients with generalised myasthenia gravis (ADAPT): a multicentre, randomised, placebo-controlled, phase 3 trial. Lancet Neurol. 2021 Jul;20(7):526-536. doi: 10.1016/S1474-4422(21)00159-9. PMID 34146511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, open-label study was a follow-on study of ARGX-113-1704 (NCT03669588) and was conducted in participants with myasthenia gravis having generalized muscle weakness at 51 investigational sites in 14 countries between 01 Mar 2019 and 30 Jun 2022. This study was conducted in 2 sequential parts: Part A (1 year) and Part B (<=2 years).
Pre-assignment Details: Participants from ARGX-113-1704 who either completed that study or required retreatment that could not be completed during a treatment cycle in that study were included in this study to receive efgartigimod. A total of 151 participants rolled over to this study and 145 of them received at least 1 dose of study treatment. Participants starting part B of this study were eligible to roll over in ARGX-113-2002 study.
Groups:
- Efgartigimod: Participants were administered efgartigimod intravenous (IV) 10 milligrams/kilograms (mg/kg) over 1 hour every 7 days for 4 administrations per treatment period (TP) for 3 weeks in this study irrespective of whether they received efgartigimod or placebo in ARGX-113-1704. After the fourth infusion, participants entered an intertreatment period (ITP) of variable duration (minimum 4 weeks between treatment periods). Subsequent TPs were implemented according to clinical response.
Period: Overall Study
Arm/Group | Efgartigimod
Started | 145
Completed | 28
Not Completed | 117
Not completed — Adverse Event | 8
Not completed — Death | 5
Not completed — Physician Decision | 1
Not completed — Sponsor decision | 1
Not completed — Study terminated by Sponsor | 1
Not completed — Withdrawal by Subject | 13
Not completed — Other | 88

BASELINE CHARACTERISTICS:
Population: The Safety Analysis set consisted of all participants who rolled over from ARGX-113-1704 and received >=1 dose or part of a dose of efgartigimod in this study.
Groups:
- Efgartigimod: Participants were administered efgartigimod IV 10 mg/kg over 1 hour every 7 days for 4 administrations per TP for 3 weeks in this study irrespective of whether they received efgartigimod or placebo in ARGX-113-1704. After the fourth infusion, participants entered an ITP of variable duration (minimum 4 weeks between treatment periods). Subsequent TPs were implemented according to clinical response.
Arm/Group | Efgartigimod
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (14.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 11
  Black or African American | 5
  White | 126
  Multiple | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 10
  Hispanic or Latino | 9
  Not Hispanic or Latino | 126
Anti-acetylcholine receptor antibodies (AChR-Ab) status [Count of Participants; unit: Participants]
  AChR-Ab seropositive | 111
  AChR-Ab seronegative | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious AEs, TEAEs Leading to Study Drug Discontinuation and Fatal TEAE in AChR-Positive Participants
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any clinically significant abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (electrocardiogram [ECG], radiological scans, vital signs measurements) were collected as AEs. All AEs starting on or after first dose administered and until completion of participant's last visit were considered as TEAEs. A serious AE (SAE) was any AE that resulted in death, was life-threatening, required inpatient hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality, or was medically significant.
Time Frame: TEAEs were collected from the start of first administered study treatment (Day 1) up to end of follow-up, approximately up to 3 years
Population: The Safety Analysis set consisted of all participants who rolled over from ARGX-113-1704 and received >=1 dose or part of a dose of efgartigimod in this study. Only those participants with AChR-positive status are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod
Number analyzed (Participants) | 111
Participants
  TEAE | 92
  Treatment-emergent SAE | 28
  TEAEs leading to study drug discontinuation | 10
  Fatal TEAE | 4

2. Secondary Outcome: Number of Participants With TEAEs, Treatment-Emergent SAEs, TEAEs Leading to Study Drug Discontinuation and Fatal TEAE in the Overall Population
Description: Overall population included both AChR-Ab seropositive and AChR-Ab seronegative participants. An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any clinically significant abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (ECG, radiological scans, vital signs measurements) were collected as AEs. All AEs starting on or after first dose administered and until completion of participant's last visit were considered as TEAEs. An SAE was any AE that resulted in death, was life-threatening, required inpatient hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality, or was medically significant.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod
Number analyzed (Participants) | 145
Participants
  TEAE | 124
  Treatment-emergent SAE | 36
  TEAEs leading to study drug discontinuation | 12
  Fatal TEAE | 5

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the start of first administered study treatment (Day 1) up to end of follow-up, approximately up to 3 years
Description: The Safety Analysis set consisted of all participants who rolled over from ARGX-113-1704 and received >=1 dose or part of a dose of efgartigimod in this study.
Arm/Group | Efgartigimod
All-Cause Mortality (participants affected / at risk) | 5/145
Serious Adverse Events (participants affected / at risk) | 36/145
Other Adverse Events (participants affected / at risk) | 83/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efgartigimod (N=145)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Defect conduction intraventricular (Cardiac disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 2 (2)
Dysentery (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia escherichia (Infections and infestations) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 7 (7)
Myasthenia gravis crisis (Nervous system disorders) | 2 (2)
Stupor (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 1 (1)
Spinal operation (Surgical and medical procedures) | 1 (1)
Shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efgartigimod (N=145)
Diarrhoea (Gastrointestinal disorders) | 13 (18)
Nausea (Gastrointestinal disorders) | 9 (13)
Pyrexia (General disorders) | 11 (11)
COVID-19 (Infections and infestations) | 16 (16)
Nasopharyngitis (Infections and infestations) | 20 (24)
Urinary tract infection (Infections and infestations) | 12 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (15)
Headache (Nervous system disorders) | 36 (103)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Hypertension (Vascular disorders) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT03770403/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT03770403/SAP_001.pdf